CLINICAL TRIAL: NCT05074953
Title: Post-COVID-19 Monitoring in Routine Health Insurance Data
Acronym: POINTED
Status: Completed | Type: Observational
Sponsor: Technische Universität Dresden (Other)
Collaborators: InGef - Institut für angewandte Gesundheitsforschung Berlin GmbH (Unknown); BARMER Institut für Gesundheitssystemforschung (bifg) (Unknown); AOK Bayern (Industry); AOK PLUS (Industry); DAK Gesundheit (Other); Techniker Krankenkasse (Other)
Responsible Party: Principal Investigator, Falko Tesch, Principal Investigator, Technische Universität Dresden
Other Study IDs: POINTED
Record Dates: First submitted 2021-10-02; First posted 2021-10-12 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-02

CONDITIONS: Virus Diseases; Epidemiology
Keywords: Post-COVID; Cohort study; Children
MeSH Terms: conditions — Virus Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Adults: 145184 patients with COVID-19 over 17 years of age.
  Interventions: Other: Exposed to a SARS-CoV-2 infection
- Children and adolescents: 11950 patients with COVID-19 under 18 years of age.
  Interventions: Other: Exposed to a SARS-CoV-2 infection

INTERVENTIONS:
Other: Exposed to a SARS-CoV-2 infection — The study compared humans exposed to the SARS-CoV-2 infection with a matched group of those not exposed. No Intervention was applied.

SUMMARY:
The SARS-CoV-2 infection was in 2020 responsible for new disease related chronic conditions which have been referred to as Post-COVID. To date it is still unknown how common this condition is and which symptoms are related to it. The aim of the study is to monitor the onset of these conditions in a large observational study consisting of German health insurance data.

DETAILED DESCRIPTION:
SARS-CoV-2 is a virus of the coronavirus family, which includes a large number of viruses that can cause a wide variety of diseases in humans. The SARS-CoV-2 virus causes acute symptoms associated with the infection and can cause chronic conditions known as Post-COVID. To understand the prevalence and variety of Post-COVID a large observational study of health insurance data from Germany was set up. The exposed patients were identified by a diagnosis indicating a confirmed laboratory test for COVID.

The basic question concerns the burden of the Post-COVID condition. The study investigate which symptoms are more common in humans after the exposure to the virus compared to a matched unexposed cohort. Further will this be investigated in the subgroup of children and adolescents and those who have been hospitalized due to the virus infection.

ELIGIBILITY:
Inclusion Criteria:

* At least one outpatient or inpatient diagnosis of COVID-19 with laboratory detection of the virus (ICD-10: U07.1!)
* Continuously insured with the respective health insurance between 2019-01-01/birth and 2020-12-31/death

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients were collected from six different health insurances in Germany during the first and second quarter in 2020. All insurances together have over 35 million members.
Sampling Method: Non-Probability Sample
Enrollment: 157134 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of abdominal pain | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of abdominal pain recorded in outpatient or inpatient setting
Incidence of acute pain | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of acute pain recorded in outpatient or inpatient setting
Incidence of adjustment disorder | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of adjustment disorder recorded in outpatient or inpatient setting
Incidence of anuria/oliguria | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of anuria/oliguria in outpatient or inpatient setting
Incidence of anxiety disorder | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of anxiety disorder in outpatient or inpatient setting
Incidence of arthritides | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of arthritides in outpatient or inpatient setting
Incidence of ascites | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of ascites in outpatient or inpatient setting
Incidence of behavioral symptoms | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of behavioral symptoms in outpatient or inpatient setting
Incidence of cachexia | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of cachexia in outpatient or inpatient setting
Incidence of carditis due to viruses | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of carditis due to viruses in outpatient or inpatient setting
Incidence of changes in bowel habits | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of changes in bowel habits due to viruses in outpatient or inpatient setting
Incidence of chronic fatigue syndrome | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of chronic fatigue syndrome in outpatient or inpatient setting
Incidence of cognitive function impairment | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of cognitive function impairment in outpatient or inpatient setting
Incidence of concentration impairment/concentration deficit | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of concentration impairment/concentration deficit in outpatient or inpatient setting
Incidence of cough | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of cough in outpatient or inpatient setting
Incidence of COVID toe | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of COVID toe in outpatient or inpatient setting
Incidence of depression | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of depression in outpatient or inpatient setting
Incidence of developmental delay | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of developmental delay in outpatient or inpatient setting
Incidence of disorientation | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of disorientation in outpatient or inpatient setting
Incidence of dysgeusia | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of dysgeusia in outpatient or inpatient setting
Incidence of dyslexia | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of dyslexia in in outpatient or inpatient setting
Incidence of dysmenorrhea | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of dysmenorrhea in outpatient or inpatient setting
Incidence of dysphagia | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of dysphagia in outpatient or inpatient setting
Incidence of dyspnea | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of dyspnea in outpatient or inpatient setting
Incidence of dysuria | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of dysuria in outpatient or inpatient setting
Incidence of emotional and behavioral disorder | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of emotional and behavioral disorder in outpatient or inpatient setting
Incidence of epistaxis | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of epistaxis in outpatient or inpatient setting
Incidence of eye pain | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of eye pain in outpatient or inpatient setting
Incidence of facial nerve paralysis | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of facial nerve paralysis in outpatient or inpatient setting
Incidence of fever | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of fever in outpatient or inpatient setting
Incidence of flatulence | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of flatulence in outpatient or inpatient setting
Incidence of gangrene | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of gangrene in outpatient or inpatient setting
Incidence of general symptoms | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of general symptoms in outpatient or inpatient setting
Incidence of hair loss | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of hair loss in outpatient or inpatient setting
Incidence of headache | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of headache in outpatient or inpatient setting
Incidence of hearing loss/tinnitus | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of hearing loss/tinnitus in outpatient or inpatient setting
Incidence of heart failure | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of heart failure in outpatient or inpatient setting
Incidence of heart murmurs | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of heart murmurs in outpatient or inpatient setting
Incidence of heartburn | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of heartburn in outpatient or inpatient setting
Incidence of hemorrhage | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of hemorrhage in outpatient or inpatient setting
Incidence of hepatomegaly and splenomegaly | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of hepatomegaly and splenomegaly in outpatient or inpatient setting
Incidence of hoarseness | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of hoarseness in outpatient or inpatient setting
Incidence of hyperhidrosis | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of hyperhidrosis in outpatient or inpatient setting
Incidence of hypotension | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of hypotension in outpatient or inpatient setting
Incidence of impaired balance | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of impaired balance in outpatient or inpatient setting
Incidence of joint pain | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of joint pain in outpatient or inpatient setting
Incidence of loss of appetite | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of Loss of appetite in outpatient or inpatient setting
Incidence of lymphadenopathy | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of lymphadenopathy in outpatient or inpatient setting
Incidence of Malaise/fatigue/exhaustion | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of Malaise/fatigue/exhaustion in outpatient or inpatient setting
Incidence of memory impairment | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of memory impairment in outpatient or inpatient setting
Incidence of meningismus | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of meningismus in outpatient or inpatient setting
Incidence of mood disorder | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of mood disorder in outpatient or inpatient setting
Incidence of movement disorders | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of movement disorders in outpatient or inpatient setting
Incidence of myalgia | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of myalgia in outpatient or inpatient setting
Incidence of myocardial infarction | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of myocardial infarction in outpatient or inpatient setting
Incidence of myocarditis | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of myocarditis in outpatient or inpatient setting
Incidence of nausea | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of nausea in outpatient or inpatient setting
Incidence of neurasthenia | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of neurasthenia in outpatient or inpatient setting
Incidence of neurological manifestation of Post-COVID | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of Neurological manifestation of Post-COVID in outpatient or inpatient setting
Incidence of obsessive-compulsive disorder | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of obsessive-compulsive disorder in outpatient or inpatient setting
Incidence of oedema | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of oedema in outpatient or inpatient setting
Incidence of other cardiac arrhythmias | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of other cardiac arrhythmias in outpatient or inpatient setting
Incidence of other coordination disorders/ataxia | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of other coordination disorders/ataxia in outpatient or inpatient setting
Incidence of other symptoms of the urinary system | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of other symptoms of the urinary system in outpatient or inpatient setting
Incidence of pain, not elsewhere classified | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of pain, not elsewhere classified in outpatient or inpatient setting
Incidence of paresis | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of paresis in outpatient or inpatient setting
Incidence of paresthesia of skin | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of paresthesia of skin in outpatient or inpatient setting
Incidence of pathological findings from male genital tract | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of pathological findings from male genital tract in outpatient or inpatient setting
Incidence of pathological lung findings | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of pathological lung findings from male genital tract in outpatient or inpatient setting
Incidence of pathological reflexes | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of pathological reflexes in outpatient or inpatient setting
Incidence of pericarditis | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of pericarditis in outpatient or inpatient setting
Incidence of polyuria | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of polyuria in outpatient or inpatient setting
Incidence of Post-COVID | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of Post-COVID in outpatient or inpatient setting
Incidence of pulmonary embolism | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of pulmonary embolism in outpatient or inpatient setting
Incidence of rash | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of rash in outpatient or inpatient setting
Incidence of respiratory insufficiency | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of respiratory insufficiency in outpatient or inpatient setting
Incidence of seizures | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of seizures in outpatient or inpatient setting
Incidence of sensation and perception disorder | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of sensation and perception disorder in outpatient or inpatient setting
Incidence of shock | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of shock in outpatient or inpatient setting
Incidence of sinus vein thrombosis | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of sinus vein thrombosis in outpatient or inpatient setting
Incidence of sleep disorders | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of sleep disorders in outpatient or inpatient setting
Incidence of somatization disorder | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of somatization disorder in outpatient or inpatient setting
Incidence of somnolence | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of somnolence in outpatient or inpatient setting
Incidence of sopor/coma | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of sopor/coma in outpatient or inpatient setting
Incidence of speech and language disorders | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of speech and language disorders in outpatient or inpatient setting
Incidence of stroke | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of stroke in outpatient or inpatient setting
Incidence of subcutaneous nodules | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of subcutaneous nodules in outpatient or inpatient setting
Incidence of syncope | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of syncope in outpatient or inpatient setting
Incidence of tetany | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of tetany in outpatient or inpatient setting
Incidence of throat/chest pain | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of throat/chest pain in outpatient or inpatient setting
Incidence of thrombosis | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of thrombosis in outpatient or inpatient setting
Incidence of urethral discharge | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of urethral discharge in outpatient or inpatient setting
Incidence of urinary retention | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of urinary retention in outpatient or inpatient setting
Incidence of vertigo | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of vertigo in outpatient or inpatient setting
Incidence of visual disturbances | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of visual disturbances in outpatient or inpatient setting
Incidence of weight gain/loss, eating disorders | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of weight gain/loss, eating disorders in outpatient or inpatient setting

CONTACTS AND LOCATIONS:
Overall Officials: Falko Tesch, Principal Investigator — Center for Evidence-Based Healthcare, Technische Universität Dresden; Jochen Schmitt, MD, MPH, Study Director — Center for Evidence-Based Healthcare, Technische Universität Dresden
Locations (1):
- Center for Evidence-Based Healthcare, Dresden, Saxony, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ehm F, Tesch F, Menzer S, Loser F, Bechmann L, Vivirito A, Wende D, Batram M, Buschmann T, Ludwig M, Roessler M, Seifert M, Sarganas Margolis G, Reitzle L, Koenig C, Schulte C, Ballesteros P, Bassler S, Bitterer T, Riederer C, Berner R, Scheidt-Nave C, Schmitt J, Toepfner N. Long/post-COVID in children and adolescents: symptom onset and recovery after one year based on healthcare records in Germany. Infection. 2025 Feb;53(1):415-426. doi: 10.1007/s15010-024-02394-8. Epub 2024 Sep 16. PMID 39285063
- [Background] Roessler M, Tesch F, Batram M, Jacob J, Loser F, Weidinger O, Wende D, Vivirito A, Toepfner N, Ehm F, Seifert M, Nagel O, Konig C, Jucknewitz R, Armann JP, Berner R, Treskova-Schwarzbach M, Hertle D, Scholz S, Stern S, Ballesteros P, Bassler S, Bertele B, Repschlager U, Richter N, Riederer C, Sobik F, Schramm A, Schulte C, Wieler L, Walker J, Scheidt-Nave C, Schmitt J. Post-COVID-19-associated morbidity in children, adolescents, and adults: A matched cohort study including more than 157,000 individuals with COVID-19 in Germany. PLoS Med. 2022 Nov 10;19(11):e1004122. doi: 10.1371/journal.pmed.1004122. eCollection 2022 Nov. PMID 36355754
- See also: Related Info — https://www.rki.de/DE/Content/InfAZ/N/Neuartiges_Coronavirus/Long-COVID/POINTED.html